CLINICAL TRIAL: NCT06175039
Title: Investigation of the Efficiency of Pulmonary Rehabilitation With Telerehabilitation Method in Patients With Bronchiectasis
Brief Title: Telerehabilitation in Patients With Bronchiectasis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Saglik Bilimleri Universitesi (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: BronsTeleReh-1
Record Dates: First submitted 2023-11-23; First posted 2023-12-18 (Actual); Last update posted 2024-06-07 (Actual); Status verified 2023-11

CONDITIONS: Bronchiectasis
Keywords: bronchiectasis; pulmonary rehabilitation; telerehabilitation
MeSH Terms: conditions — Bronchiectasis

STUDY DESIGN:
Intervention Model Description: The cases meeting the inclusion criteria will be randomized and divided into two groups, the groups will be named as Telerehabilitation Exercise Group (TRGr) and Control Group (KGr).
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Telerehabilitation Exercise Group (Experimental)
  Interventions: Other: Telerehabilitation exercise program
- Control Group (Other)
  Interventions: Other: Control program

INTERVENTIONS:
Other: Telerehabilitation exercise program — TRGr will be given online exercises, synchronized 3 days a week, accompanied by a physiotherapist, via videoconference on the group smartphone.
  Arms: Telerehabilitation Exercise Group
Other: Control program — KGr will be a pulmonary rehabilitation information brochure will be given after the initial evaluation. They will be asked to do the exercises on the brochure.
  Arms: Control Group

SUMMARY:
It is to determine the effectiveness of pulmonary rehabilitation by telerehabilitation method in bronchiectasis patients. The cases meeting the inclusion criteria will be randomized and divided into two groups, the groups will be named as Telerehabilitation Exercise Group (TRGr) and Control Group (CGr).

DETAILED DESCRIPTION:
Patients diagnosed with bronchiectasis by HRCT by a chest diseases specialist and referred to pulmonary rehabilitation by determining the severity of bronchiectasis with the Modified Reiff Score and Bronchiectasis Severity Index Score will be included in the study.

The cases meeting the inclusion criteria will be randomized and divided into two groups, the groups will be named as Telerehabilitation Exercise Group (TRGr) and Control Group (KGr). TRGr will be given online exercises, synchronized 3 days a week, accompanied by a physiotherapist, via videoconference on the group smartphone. As for the KGr group, a pulmonary rehabilitation information brochure will be given to after the initial evaluation. They will be asked to do the exercises on the brochure. The exercise period will be 8 weeks for both groups. Standard medical treatments for both groups will continue.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 and over
* Diagnosed with bronchiectasis by HRCT
* Stable clinical state at the time of admission without infection or exacerbation in the previous 3 weeks
* Know how to use technological devices

Exclusion Criteria:

* A history of effort-related syncope or any comorbidity (such as severe orthopedic or neurological deficits or unstable heart disease) that precludes exercise training
* Patients with systemic diseases other than bronchiectasis that also affect the lungs, such as systemic lupus erythematosus, infection, interstitial lung disease, lung cancer, heart and kidney failure, which will cause shortness of breath
* Having balance problems that prevent them from doing exercises
* Participation in a pulmonary rehabilitation program within the past 12 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2023-05-15 (Actual); Primary Completion 2024-03-16 (Actual); Study Completion 2024-06-04 (Actual)

PRIMARY OUTCOMES:
The exercise capacity | Change from baseline incremental shuttle walking distance at 8 weeks
  The exercise capacity will be assessed by the incremental shuttle walking test.

SECONDARY OUTCOMES:
Forced vital capacity (FVC) | Change from baseline FVC at 8 weeks
  Forced vital capacity will be assessed by the spirometer. Pulmonary function test will performe by using the Pony Fx spirometry device, and according to the American Thoracic Society (ATS) guidelines
Forced expiratory volume in one second (FEV1) | Change from baseline FEV1 at 8 weeks
  Forced expiratory volume in one second will be assessed by the spirometer. Pulmonary function test will performe by using the Pony Fx spirometry device, and according to the American Thoracic Society (ATS) guidelines
Respiratory muscle strength | Change from baseline respiratory muscle strength at 8 weeks
  Respiratory muscle strength will be evaluated by the intraoral pressure measurement device.The mouth pressure measurement was performed with the Cosmed Pony Fx. Patient placed a rubber mouthpiece with flanges, on the device, sealed their lips firmly around the mouthpiece, exhaled/inhaled slowly and completely, and then tried to breath in as hard as possible. The patient was allowed to rest for about a minute and the maneuver was repeated five times. Verbal or visual feedback was provided after each maneuver. The aim is that the variability between measurements is less than 10 cm H2O. The maximum value was obtained.
Peripheral muscle strength | Change from baseline peripheral muscle strength at 8 weeks
  Peripheral muscle strength will be assessed by the hand held dynamometer
Perception of dyspnea | Change from baseline dyspnea perception at 8 weeks
  Perception of dyspnea will be evaluated by Modified Medical Research Council Dyspnea scale. The mMRC Dyspnea Scale is best used to establish baseline functional impairment due to dyspnea attributable to respiratory disease; tracking the mMRC over time or with therapeutic interventions is of less certain clinical utility.The severity of dyspnea is rated on a scale of 0 to 4. "O" means no dyspnea perception, "4" means severe dyspnea perception.
Saint George Respiratory Questionnaire (SGRQ) score | Change from baseline SGRQ score at 8 weeks
  The quality of life will be assessed by the Saint George Respiratory Questionnaire.The SGRQ ranges from 0 (no impairment of quality of life) to 100 (highest impairment of quality of life)
Modified Borg Scale | Change from baseline Modified Borg Scale score at 8 weeks
  Exertion and rest define the level of dyspnea. It consists of ten items that describe the severity of dyspnea according to its degree. A minimum of 1 and a maximum of 10 points can be obtained. 1, no shortness of breath. 10, maximal shortness of breath.
Leicester Cough Questıonnaıre (LCQ) | Change from baseline LCQ score at 8 weeks
  The cough will be assessed by the Leicester Cough Questionnaire. It includes physical, psychological and social sub-parameters and each item is scored between 1-7. High scores indicate that the cough is less affected, while low scores indicate that the cough is more affected.

CONTACTS AND LOCATIONS:
Overall Officials: Esra Pehlivan, Assoc.Prof.Dr., Principal Investigator — Advisor; Busra Ocal, Master Degree Student, Study Chair — Student
Locations (1):
- Saglik Bilimleri University, Istanbul, Uskudar, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No